CLINICAL TRIAL: NCT05662709
Title: Leukocyte and Platelet-rich Fibrin (L-PRF) Effects on Alveolar Ridge Preservation. A Randomized Controlled Clinical Trial With One Year Follow up
Brief Title: Leukocyte and Platelet-rich Fibrin (L-PRF) Effects on Alveolar Ridge Preservation. A Randomized Controlled Clinical Trial.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, Carolina Encalada Abad, DDS, PhD candidate, Master in Periodontology and Implant dentistry., Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17/262-O_P
Record Dates: First submitted 2022-12-07; First posted 2022-12-22 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Alveolar Ridge Preservation; Dental Implants
Keywords: platelet-rich fibrin; bone regeneration; alveolar ridge preservation; tooth extraction
MeSH Terms: interventions — Tooth Extraction

STUDY DESIGN:
Intervention Model Description: Controlled clinical trial, 2 groups of patients undergoing tooth extraction, allocated to:
  * Test group: alveolar ridge preservation with L-PRF
  * Control group: spontaneous healing of the socket
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor blinded for treatment groups.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- L-PRF (Experimental): Test group, alveolar ridge preservation with L-PRF after tooth extraction.
  Interventions: Procedure: Tooth extraction; Procedure: Alveolar ridge preservation with L-PRF
- Spontaneous Healing (SH) (No Intervention): Control group, spontaneous healing of the socket after tooth extraction

INTERVENTIONS:
Procedure: Tooth extraction — Tooth extraction in the most atraumatic way
  Arms: L-PRF
Procedure: Alveolar ridge preservation with L-PRF — Blood will be drawn from the patient, centrifugued and leukocyte and platelet-rich fibrin (L-PRF) will be obtained. L-PRF plugs and membranes will be prepared and placed in the socket after extraction
  Arms: L-PRF

SUMMARY:
The goal of this clínical trial is to compare in patients needing extraction of anterior teeth the effects of leukocyte-and platelet-rich fibrin (L-PRF) for alveolar ridge preservation versus spontaneous healing. The main questions it aims to answer are:

* Does L-PRF use as alveolar ridge preservation material diminish volumetric changes in the alveolar ridge produced after tooth extraction and further bone regeneration needs?
* Does it have any advantage for wound healing and patient-related outcomes? Participants will undergo
* Tooth extraction
* Alveolar ridge preservation/ spontaneous healing
* Implant placement

Researchers will compare alveolar ridge preservation with L-PRF with spontaneous healing to see if there is an effect on reducing ridge dimensional changes happening after tooth extraction.

DETAILED DESCRIPTION:
-Objectives

The main objective is to determine if L-PRF use as alveolar ridge preservation material diminishes volumetric changes in the alveolar ridge produced after tooth extraction and needs of bone regeneration previous or simultaneous to implant placement compared to spontaneous healing.

Secondary objectives:

To determine if there are differences in wound healing after the use of L-PRF compared to spontaneous healing.

To investigate if there are differences in Patient Reported Outcome measures after the use of L-PRF compared to spontaneous healing.

To analyse the histologic differences in quality of bone after the use of L-PRF compared to spontaneous healing.

-Material and Methods

Randomized clinical trial developed in an academic onset, parallel groups, single-blinded with one year follow up after implant loading.

Ethical Aspects:

This investigation will be based on compliance with the principles of the Declaration of Helsinki. The ethics committee of Hospital Clínico San Carlos will be in charge of evaluating and approving this protocol. All patients will be fully informed before their inclusion in the study by means of informed consent.

Treatment:

All the participants will be treated by postgraduate students at the Master of Periodontology and Implant dentistry from the Complutense University of Madrid.

Twenty-eight patients in need of extraction will be included in the study. In the baseline visit local anesthesia will be administered and tooth extraction will be performed in the least traumatic way possible. The group will be allocated according to a computer-generated randomization list and given in a sealed envelope. For the test group (L-PRF) venipuncture (median basilica vein, median cubital vein, median cephalic vein) will be performed by a nurse and blood will be drawn into 8 sterile plastic 10 ml tubes without anticoagulant (Vacutainers: IntraSpin™, Intra-lock,USA). L-PRF plugs and membranes will be prepared as described by Choukroun et al 2001. Tubes will be centrifuged for 12 minutes at 2700 rpm using a table centrifuge (IntraSpin™, IntraLock, USA). After centrifugation, clots will be removed from the tubes, separated from red element phase at the base with pliers and placed in a metal tray (Xpression™ Box). Four to five of them will be packed in a cylinder to obtain plugs, and four will be squeezed between the tray and a glass plate to obtain L-PRF membranes. In sockets of the L-PRF group, 2-5 plugs, depending on the size of the socket will be inserted and compressed and membranes will be adapted on top and inserted in vestibular and lingual envelope flaps previously prepared. A crossed horizontal mattress suture (Polyamide 5.0, Supramid™, SMI AG, Steinerberg, Belgium) will be placed on top. In the control group, after extraction, just the suture will be performed to stabilize the coagulum. Patients will be prescribed ibuprofen (600mg t.i.d) or paracetamol (1g t.i.d) and chlorhexidine 0.12% + 0.05% CPC mouth rinse (PerioAid® Tratamiento, Dentaid, Barcelona, Spain) for one week.

Follow up visits:

After extraction, a cone-beam computed tomography (CBCT) scan (i-CAT Classic, Imaging Sciences International, Hatfield, Pennsylvania) and a digital impression (Medit i500 ™, Medit, Seoul, Korea) to obtain a stereolithographic model of the area will be taken.

Sutures will be removed at 7days. Patients will attend follow-up visits at 4 weeks and 4 months to monitor wound healing. Patient reported outcome measures (PROM's) will be registered at 1 and 4 weeks.

Diagnostic for implant placement:

Four months after tooth extraction, the new CBCT will be assessed to see bone availability for implant placement. In this visit a new digital impression will be taken to assess dimensional changes in bone and soft tissue with an image analysis software (SMOP®, Swissmeda, Switzerland).

Implant surgery will be scheduled, it will be determined if bone regeneration is necessary before or simultaneously to implant placement. At the time of implant placement, a biopsy will be taken for histologic analysis with a trephine bur of 2.5mm diameter (Komet, USA) with the aim to obtain a sample of healed bone tissue and perform histologic analysis. After osteotomy, an implant Gold & Blue (Intralock, USA) will be inserted. If there is no need of bone regeneration, healing abutments will be placed; if there is need of simultaneous bone regeneration the width and height of the defect will be registered and a bone substitute NanoBone®(Intra-lock Iberia, Madrid Spain) and a resorbable collagen membrane (Bio-Gide; Geistlich, Switzerland will be placed, with a submerged healing protocol. Four months late, second stage surgery will be performed. If implant cannot be properly stabilized, a guided bone regeneration will be performed with the same materials and implants will be placed after six months.

After implant placement, a periapical x-ray will be performed, and sutures will be removed after one week.

Implant restoration:

After a healing period of 10 weeks after implant placement (between 4-6 months if bone regeneration has been required), impressions will be taken to make the provisional or final prosthesis, STLs models for ridge changes assessment and implant related variables will be registered.

The day of implant loading, a new standardized periapical x-ray will be taken with a personalized bite block. Peri-implant health related variables will be assessed, and esthetic outcomes will be registered. This will be the baseline visit for the follow up analysis of the implants placed.

Implants follow up:

The implants will be assessed at 6 and 12 months after loading the final prosthesis. In these visits, the same clinical variables related to peri-implant health and aesthetics will be recorded as in the baseline visit (definitive load). Additionally, at 12 months a periapical X-ray will be performed, a digital impression of the treated area will be taken and a satisfaction questionnaire will be given to the patient.

-Sample size calculation

The sample size calculation was based on detecting a mean difference in reduction of the HRW of 2,3mm with an estimated standard deviation (SD) of 1.1 between groups (Thalmair et al., 2013). To detect statistically significant differences (α=0.05) with a 90% power, a minimum of 11 subjects per group are needed, which including an expected 20% drop-out rate, it resuls in a final sample of 14 participants per group.

-Data analysis

Data will be analyzed to compare both treatment modalities. The normality of the distribution will be evaluated using the Kolmogorov-Smirnov test. Depending on the distribution of the data, parametric or non-parametric tests will be used. Quantitative variables will be assessed by means of student´s t test or Mann Whitney´s U test.

Qualitative variables will be expressed through distribution frequencies and will be compared with chi-square tests.

The clinical significance level is set at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy patients ≥18 years old
* Need for extraction of a tooth in the anterior area (position of second premolar to second premolar in maxilla or mandible) that needs to be replaced by an implant-supported restoration
* Presence of natural teeth mesially and distally of tooth to be extracted, periodontally healthy (probing depths <5 mm without bleeding on probing).

Exclusion Criteria:

* Systemic conditions affecting bone or soft tissue healing
* Smokers of more than 10 cigarettes a day or equivalent to cigarettes
* Breastfeeding or pregnant women
* Patients without availability to attend follow-up visits or patients rejecting to sign the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
Radiographic linear changes in horizontal width of the alveolar ridge | From tooth extraction (Baseline) to four months healing (4m)
  Cuantitative variable. A validated method to superimpose the radiographs will be used (Ortiz-Vigón et al., 2018; Sanz-Martín et al., 2019).A digital imaging software (SMOP®, Swissmeda Ltd©, Zurich, Switzerland) is used to convert DICOM files into STL files. The images from Baseline and 4 months CBCTs were superimposed using common reference points. After a "fine fit" of the two surfaces, it will appear as a merged contour in axial, coronal, and sagittal views. The center of the alveolus will be determined mesiodistally in the occlusal view. Linear changes in width between 4 months and baseline will be determined by horizontal lines drawn perpendicular to the longitudinal axis in the center of the socket. Three measurements will be taken at 1mm (HRW1), 3mm (HRW3), and 5mm (HRW5) below the Bl bone crest. The change will be calculated by subtraction of the 4 months to Baseline distance in millimeters.

SECONDARY OUTCOMES:
Radiographic linear changes height of the alveolar ridge | From tooth extraction (Baseline) to four months healing (4m)
  Cuantitative variable. A validated method to superimpose the radiographs will be used (Ortiz-Vigón et al., 2018; Sanz-Martín et al., 2019).A digital imaging software (SMOP®, Swissmeda Ltd©, Zurich, Switzerland) is used to convert DICOM files into STL files. The images from Baseline and 4 months CBCTs were superimposed using common reference points. After a "fine fit" of the two surfaces, it will appear as a merged contour in axial, coronal, and sagittal views. The center of the alveolus will be determined mesiodistally in the occlusal view. Vertical changes will be determined by measuring the distance from the most coronal aspect of the crest at 4 months to the crest at baseline at buccal and lingual aspects.
Changes in ridge contour | From tooth extraction (Baseline) to four months healing (4m)
  Cuantitative variable . A similar superimposition method will be used for ridge contour analysis in STL files (Bienz et al., 2017). An image analysis software (SMOP®, Swissmeda, Sweden) will be used to superimpose STL files taken after tooth extraction and at 4 months. Horizontal lines will be drawn perpendicular to the longitudinal axis in the center of the socket at 1mm, 3mm, and 5mm below the crestal margin. Dimensional changes will be calculated by subtraction of the 4 months to baseline distances in millimeters. Vertical changes will be registered as the distance between contours of both time points in the center of the alveolus.
Volumetric changes | From tooth extraction (Baseline) to four months healing (4m)
  Cuantitative variable. Changes in volume of a region of interest (ROI) delimited by the crestal margin, the mesial and distal line angles of adjacent teeth, and extending 5 mm apically will be calculated in the superimposed images by the software (SMOP®, Swissmeda, Sweden)
Patient reported outcome measures | At one week, one month and four months visit.
  Cuantitative variable. Patients perception of pain, inflammation, bleeding and functional capacity reported in a VISUAL ANALOGUE (VAS) scale, with scores fro 0-10.
  Regarding inflammation, pain and bleeding lower scores will mean better performance of intervention and higher outcomes worse performance.
  Regarding functional capacity, higher scores will mean better performance and lower scores will mean worse performance.
Bone regeneration needs | 4 months after tooth extraction
  Cualitative variable. At the moment of implant planning, bone availability will be assessed and it will be determined if there is a need of bone regeneration previous or simultaneous to implant placement
Percentage of mineralized bone | 4 months after tooth extraction, during the implant placement surgery.
  Cuantitative variable. Histological analysis. Assessment of the percentage of mineralized bone in the core biopsies taken at implant placement.

OTHER OUTCOMES:
Peri implant probing depth | At implant placement, 6 months and 12 months after loading
  Cuantitative variable: Probing depth (PD). Distance in millimeters m from the bottom of the pocket to the gingival margin.
Peri-implant Plaque index | At implant placement, 6 months and 12 months after loading
  Cualitative variable: Presence or absence (yes/no) of plaque around 6 points of the implant site. Mesiobuccal, Midbuccal, Distobuccal; Mesiolingual, Midlingual, Distolingual
Bleeding on probing | At implant placement, 6 months and 12 months after loading
  Cualitative variable: Presence or absence (yes/no) of bleeding after probing in 6 points around the implant site. Mesiobuccal, Midbuccal, Distobuccal; Mesiolingual, Midlingual, Distolingual.
Radiographic changes in bone levels | At implant placement, 6 months and 12 months after loading
  An analysis of periapical radiographs will be performed to assess changes in bone levels at 12 months after loading. Defined as the distance between the implant shoulder and the first bone-to-implant contact a mesial and distal aspects
Clinical crown dimension | At implant loading, 6 months and 12 months follow up
  Distance in millimeters from the gingival margin to the incisal edge or occlusal surface. An increase in the value would indicate a recession of the peri-implant mucosa.
Pink Esthetic Score | At implant loading, 6 months and 12 months follow up
  Pink esthetic index. According to the parameters described by (Furhäuser et al 2005), seven variables are measured to assess the status of the peri-implant soft tissues, among them: mesial papilla, distal papilla, gingival margin level, soft tissue contour, alveolar process, and tissue color and texture.
  This index is determined by granting a value of 0, 1 or 2, and combine to give a final score, the maximum final score is 14 points. Scores > or = to 12 mean high esthetic achievement.
Changes in ridge contour after loading | 12 months after implant loading
  Cuantitative variable. An image analysis software (SMOP®, Swissmeda, Sweden) will be used to superimpose stl files taken after tooth extraction and 12 months after implant loading. In a sagittal section of the superimposed images linear measurements will be taken to determine horizontal, vertical and volumetric changes.

CONTACTS AND LOCATIONS:
Locations (1):
- Complutense University of Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Choukroun, J., Adda, F., Schoeffler, C., & Vervelle, A. (2001). The opportunity in perio-implantology: The PRF. Implantodontie, 42, 55-62.
- [Background] Dohan Ehrenfest DM, de Peppo GM, Doglioli P, Sammartino G. Slow release of growth factors and thrombospondin-1 in Choukroun's platelet-rich fibrin (PRF): a gold standard to achieve for all surgical platelet concentrates technologies. Growth Factors. 2009 Feb;27(1):63-9. doi: 10.1080/08977190802636713. PMID 19089687
- [Background] Tan WL, Wong TL, Wong MC, Lang NP. A systematic review of post-extractional alveolar hard and soft tissue dimensional changes in humans. Clin Oral Implants Res. 2012 Feb;23 Suppl 5:1-21. doi: 10.1111/j.1600-0501.2011.02375.x. PMID 22211303
- [Background] Barone A, Aldini NN, Fini M, Giardino R, Calvo Guirado JL, Covani U. Xenograft versus extraction alone for ridge preservation after tooth removal: a clinical and histomorphometric study. J Periodontol. 2008 Aug;79(8):1370-7. doi: 10.1902/jop.2008.070628. PMID 18672985
- [Background] Schropp L, Wenzel A, Kostopoulos L, Karring T. Bone healing and soft tissue contour changes following single-tooth extraction: a clinical and radiographic 12-month prospective study. Int J Periodontics Restorative Dent. 2003 Aug;23(4):313-23. PMID 12956475
- [Background] Sanz-Martin I, Permuy M, Vignoletti F, Nunez J, Munoz F, Sanz M. A novel methodological approach using superimposed Micro-CT and STL images to analyze hard and soft tissue volume in immediate and delayed implants with different cervical designs. Clin Oral Implants Res. 2018 Oct;29(10):986-995. doi: 10.1111/clr.13365. Epub 2018 Sep 23. PMID 30246362
- [Background] Vignoletti F, Matesanz P, Rodrigo D, Figuero E, Martin C, Sanz M. Surgical protocols for ridge preservation after tooth extraction. A systematic review. Clin Oral Implants Res. 2012 Feb;23 Suppl 5:22-38. doi: 10.1111/j.1600-0501.2011.02331.x. PMID 22211304
- [Background] Furhauser R, Florescu D, Benesch T, Haas R, Mailath G, Watzek G. Evaluation of soft tissue around single-tooth implant crowns: the pink esthetic score. Clin Oral Implants Res. 2005 Dec;16(6):639-44. doi: 10.1111/j.1600-0501.2005.01193.x. PMID 16307569
- [Background] Ortiz-Vigon A, Suarez I, Martinez-Villa S, Sanz-Martin I, Bollain J, Sanz M. Safety and performance of a novel collagenated xenogeneic bone block for lateral alveolar crest augmentation for staged implant placement. Clin Oral Implants Res. 2018 Jan;29(1):36-45. doi: 10.1111/clr.13036. Epub 2017 Jul 14. PMID 28710793
- [Result] Anwandter A, Bohmann S, Nally M, Castro AB, Quirynen M, Pinto N. Dimensional changes of the post extraction alveolar ridge, preserved with Leukocyte- and Platelet Rich Fibrin: A clinical pilot study. J Dent. 2016 Sep;52:23-9. doi: 10.1016/j.jdent.2016.06.005. Epub 2016 Jun 20. PMID 27338946
- [Result] Temmerman A, Vandessel J, Castro A, Jacobs R, Teughels W, Pinto N, Quirynen M. The use of leucocyte and platelet-rich fibrin in socket management and ridge preservation: a split-mouth, randomized, controlled clinical trial. J Clin Periodontol. 2016 Nov;43(11):990-999. doi: 10.1111/jcpe.12612. Epub 2016 Sep 21. PMID 27509214
- [Result] Thalmair T, Fickl S, Schneider D, Hinze M, Wachtel H. Dimensional alterations of extraction sites after different alveolar ridge preservation techniques - a volumetric study. J Clin Periodontol. 2013 Jul;40(7):721-7. doi: 10.1111/jcpe.12111. Epub 2013 May 5. PMID 23647007
- [Result] Suttapreyasri S, Leepong N. Influence of platelet-rich fibrin on alveolar ridge preservation. J Craniofac Surg. 2013 Jul;24(4):1088-94. doi: 10.1097/SCS.0b013e31828b6dc3. PMID 23851746